CLINICAL TRIAL: NCT01091935
Title: Safety of Intravenous Lidocaine Infusions for Chronic Neuropathic Pain
Brief Title: Safety of Intravenous Lidocaine Infusions
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Patricia Morley-Forster, St Joseph's Health Care
Other Study IDs: R-08-341; 15240E (Other: REB)
Record Dates: First submitted 2010-03-22; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Neuropathic Pain
Keywords: Lidocaine,Intravenous Infusions,Neuropathic Pain,Side Effects
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lidocaine: Adults >18 yrs , attending St Joseph's Health Care Pain Clinic with a diagnosis of chronic neuropathic pain who are being treated with an lidocaine infusion of 5 mg/kg over 45 minutes
  Consecutive patients from two time periods:
  1. June 15 to August 21, 2009
  2. October 15-Dec 22,2009

SUMMARY:
The purpose of this study is to prospectively determine the side effects profile in adults with neuropathic pain receiving intravenous infusions of lidocaine 5 mg per kg of lean body weight, infused over 45 minutes.

DETAILED DESCRIPTION:
Eligibility Criteria:

Adults > 18 yrs with chronic central or peripheral neuropathic pain at the St Joseph's Health Care Pain Clinic between June and December 2009.

Outcome measures: All side effects spontaneously reported. Sedation, nausea, dizziness by Visual Analog Score Q 15 minutes; hemodynamic data q 5 minutes during and after infusion for 30 minutes.

Daily diary of side effects and Visual Analogue score of Pain for 7 days post-infusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients > 18 years < 80 years diagnosed with chronic neuropathic pain

Exclusion Criteria:

* Unable to provide informed consent
* Unable to speak and understand English
* Liver, kidney, or cardiac failure
* Allergy to Lidocaine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult outpatients attending St Joseph's Chronic Pain Clinic in one of two time periods who have been diagnosed with chronic neuropathic pain by clinical history and examination and are scheduled to receive a lidocaine infusion for pain management
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia K Morley-Forster, MD, FRCPC, Principal Investigator — Associate Professor,Dept of Anesthesia and Perioperative Medicine,University of Western Ontario, Lawson Health Research Institute; Patricia K Morley-Forster, MD, FRCPC, Principal Investigator — Associate Professor, University of Western Ontario, Lawson Health Research Institute
Locations (1):
- St Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Background] Attal N, Gaude V, Brasseur L, Dupuy M, Guirimand F, Parker F, Bouhassira D. Intravenous lidocaine in central pain: a double-blind, placebo-controlled, psychophysical study. Neurology. 2000 Feb 8;54(3):564-74. doi: 10.1212/wnl.54.3.564. PMID 10680784